CLINICAL TRIAL: NCT01437982
Title: A Post Marketing Surveillance to Evaluate the Safety and Efficacy of Lotemax Ophthalmic Suspension 0.5%
Brief Title: A Study to Evaluate the Safety and Efficacy of Lotemax Ophthalmic Suspension 0.5%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 628
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Conjunctivitis, Seasonal Allergic; Conjunctivitis, Giant Papillary; Inflammation
Keywords: post-operative inflammation; conjunctivitis; safety; Seasonal allergic conjunctivitis; Giant papillary conjunctivitis
MeSH Terms: conditions — Conjunctivitis; Conjunctivitis, Allergic; Inflammation | interventions — Loteprednol Etabonate; prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol Etabonate (Experimental): Ophthalmic Gel 0.5%
  Interventions: Drug: Loteprednol Etabonate
- Prednisolone Acetate 1% Oph Susp (Experimental): Ophthalmic suspension 0.5%
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp

INTERVENTIONS:
Drug: Loteprednol Etabonate — Ocular administration of study drug. at least once within any indication of the label.
  Other Names: Lotemax
  Arms: Loteprednol Etabonate
Drug: Prednisolone Acetate 1% Oph Susp — Ocular administration of study drug. at least once within any indication of the label.
  Other Names: Prednisolone Acetate
  Arms: Prednisolone Acetate 1% Oph Susp

SUMMARY:
The objective of this study is to identify any adverse events or adverse drug reactions through post-marketing surveillance under routine clinical practice

DETAILED DESCRIPTION:
The objective of this study is to identify any adverse events or adverse drug reactions through post-marketing surveillance under routine clinical practice after marketing authorization of Lotemax ophthalmic suspension 0.5%

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been treated with the study drug at least once and completed safety follow-up.
* Subjects who have been treated with the study drug at least once and completed the clinical efficacy assessment.

Exclusion Criteria:

* Subjects not treated with study drug at least once.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-08-05 (Actual); Primary Completion 2015-10-19 (Actual); Study Completion 2015-10-19 (Actual)

PRIMARY OUTCOMES:
Safety | 4 years
  All adverse events that occurred from the first dose of the study drug regardless of causality to the study drug. Changes in all undesirable medical findings and all adverse events occurring with the use of the study drug.

SECONDARY OUTCOMES:
Seasonal Allergic Conjunctivitis | 4 years
  Signs and symptoms of seasonal allergic conjunctivitis: The efficacy assessment will be evaluated according to the classification: improved, unchanged, worsened, impossible to assess.
Giant Papillary Conjunctivitis | 4 years
  Signs and symptoms of giant papillary conjunctivitis: The results of the efficacy assessment will be evaluated according to the classification: improved, unchanged, worsened, impossible to assess.
Post-operative inflammation | 4 years
  Treatment of post-operative inflammation following ocular surgery: The results of the final efficacy assessment will be evaluated according to the classification: improved, unchanged, worsened, impossible to assess.

CONTACTS AND LOCATIONS:
Overall Officials: Binu Alexander, MD, Study Director — Valeant Pharmaceuticals
Locations (1):
- Bausch & Lomb Korea Ltd, Seoul, South Korea